CLINICAL TRIAL: NCT03541395
Title: Testosterone-Dependent Effects on Protein Biomarkers From Healthy Males Before and After Pharmacological Castration
Brief Title: Testosterone-Dependent Effects on Protein Biomarkers From Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Johan Malm, Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TP 001
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testosterone (Other): A Gonadotropin releasing hormone agonist (GnRH-agonist) is administered to lower the testosterone to castration levels. After four weeks testosterone undecanoate is administered to increase the testosterone to normal levels.
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: GnRH antagonist

SUMMARY:
The study is designed to identify and validate new protein biomarkers in blood related to testosterone activity. Thirty healthy young males underwent pharmaceutical castration to lower testosterone levels. After three weeks the subjects received an intramuscular injection of testosterone undecanoate. Blood samples from just before pharmaceutical castration, three weeks after castration, and one week after injection of testosterone undecanoate were collected representing normal testosterone levels, low testosterone levels, and testosterone at eugonadal levels.

ELIGIBILITY:
Inclusion Criteria:

healthy males

Exclusion Criteria:

use of anabolic steroids, use of narcotics,

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Protein biomarkers | 48 months
  Finding new protein biomarkers related to testosterone response

CONTACTS AND LOCATIONS:
Overall Officials: Johan Malm, MD, Study Chair — Lund University; Roger Appelqvist, PhD, Principal Investigator — Lund University; Gyorgy Marko-Varga, PhD, Principal Investigator — Lund University; Aleksander Giwercman, MD, Principal Investigator — Lund University; Barbara Sahlin, MSc, Principal Investigator — Lund University